CLINICAL TRIAL: NCT07349355
Title: The Effect of In-Situ Simulation and Standardized Patient Practice on Medical Error Tendencies and Attitudes of Senior Nursing Students
Brief Title: Simulation Practices and Medical Error Tendencies in Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selçuk Görücü (Other)
Responsible Party: Sponsor-Investigator, Selçuk Görücü, Lecturer, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/024
Record Dates: First submitted 2025-11-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Patient Safety
Keywords: In-situ simulation; standardized patient; nursing students; randomized controlled trial; nursing education; medical error

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 receives training in a simulation laboratory environment using standard patient interventions.
  Interventions: Other: Standardized patient
- Group 2 (Experimental): Group 2 receives training in a real hospital setting through on-site simulations and standardized patient interventions.
  Interventions: Other: İn-situ simulation
- Group 3 (No Intervention): Group 3 is the control group. They receive traditional classroom-based theoretical instruction.

INTERVENTIONS:
Other: Standardized patient — Group 1 receives training in a simulation laboratory environment using standard patient interventions.
  Arms: Group 1
Other: İn-situ simulation — Group 2 receives training in a real hospital setting through on-site simulations and standardized patient interventions.
  Arms: Group 2

SUMMARY:
As the professional group that has the most frequent contact with patients, nurses are critical to the sustainability of safe care. Literature demonstrates that nursing practice is prone to error due to heavy workloads, time pressures, complex clinical tasks, inadequate rest, inappropriate working conditions, and the physiological strain of demanding shifts. When these conditions strain both physical and cognitive resources, the risk of errors during treatment administration increases.

Medical errors remain one of the most devastating realities of healthcare. Data from the World Health Organization reveals the significant morbidity and mortality caused by errors on a global scale. Numerous studies have demonstrated that student nurses have a significant rate of errors, and those with limited clinical experience are particularly at risk in fundamental areas such as medication administration, asepsis, and patient identification. Increasing patient numbers, short stays, rapid turnover, and the intense pace of clinics negatively impact student nurses' ability to provide safe care, prompting both educators and students to seek stronger pedagogical solutions.

This is where simulation-based training comes into play. Simulation is emerging as a contemporary teaching approach that enables students to develop their clinical skills, communication, decision-making, and self-efficacy in a risk-free, safe, and structured environment. It is increasingly being used because it supports knowledge and skill transfer, reduces fear and anxiety, strengthens self-confidence, and provides the opportunity to experience errors. In-situ simulation and standardized patient practice offer strong potential for reducing students' error proneness by providing an experience closest to real-world clinical situations. However, the lack of a study in the literature examining the effects of these two methods, particularly on the medical error proneness and attitudes of final-year nursing students, is a significant gap.

This study aims to strengthen a critical area of nursing education. The aim is to evaluate the impact of in-situ simulation and standardized patient practice on final-year nursing students' medical error proneness and attitudes toward medical errors and to reveal how they transform students' competencies in providing safe care.

ELIGIBILITY:
Inclusion Criteria: Students were included in the study if they were:

* A senior nursing student at Aydın Adnan Menderes University Faculty of Nursing
* Volunteering to participate in the study
* Not absent at any time during the study period
* Working/not working as a nurse

Exclusion Criteria:

* Graduated from a health vocational high school
* Admitted through the Foreign Student Exam (YÖS)
* Graduated from a health-related associate's degree program and then enrolled in the nursing department through the Vertical Transfer Exam (DGS)
* Students who did not wish to participate in the study were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Medical error tendency scale scores of final-year nursing students | From registration to week 8 of intervention
  Medical Error Tendency Scale
  The minimum possible score is 1, and the maximum is 5. While the scale does not have a cutoff point, an increase in the mean score indicates a low tendency for the nurse to make medical errors, while a decrease in the mean score indicates a high tendency to make errors.

SECONDARY OUTCOMES:
Medical error attitude scale scores of final year nursing students | From registration to week 8 of intervention
  Medical Error Attitude Scale
  The total scale score is calculated by dividing the total score by the number of items. The cutoff point is set at 3. Healthcare personnel scoring below 3 on the scale are considered incompetent.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study does not plan to share raw data at the individual level. However, to promote transparency of research findings, summary data (demographic characteristics, pretest and posttest scores, group comparisons, and analysis results) that do not include participant identification will be shared with researchers upon request. No personal identifying information (name, contact information, institutional information, etc.) will be shared.
Supporting Information: SAP, ICF, CSR
Time Frame: August 2026-December 2026
Access Criteria: Access to data will be available only after a written request from the researcher and a review by the research team for scientific relevance. Access will only be provided by securely transmitting designated datasets via email; no sharing will be made via any open-access repository or online platform.